CLINICAL TRIAL: NCT03454945
Title: Efficacy of Doxycycline in the Treatment of Early Stages of Mycosis Fungoides: A Randomized Controlled Trial
Brief Title: Efficacy of Doxycycline in the Treatment of Early Stages of Mycosis Fungoides
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar El Sayed, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: doxycycline
Record Dates: First submitted 2017-09-05; First posted 2018-03-06 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Lymphoma
Keywords: Mycosis fungoides; Doxycycline
MeSH Terms: conditions — Lymphoma; Mycosis Fungoides | interventions — Doxycycline; Phototherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doxycyline (Experimental): Oral Vibramycin antibiotic100 mg capsule every 12 hours for 3 months
  Interventions: Drug: Vibramycin; Device: Phototherapy
- Phototherapy (Active Comparator): UVA+ psoralen 3 sessions per week for 3 months
  Interventions: Drug: Vibramycin; Device: Phototherapy

INTERVENTIONS:
Drug: Vibramycin — Antibiotic
  Other Names: Doxy
Device: Phototherapy — UVA+Psoralen

SUMMARY:
Current study aims at assessing the efficacy of doxycycline as a potential treatment modality for early stages of MF.

DETAILED DESCRIPTION:
Objectives

Objective is to evaluate the efficacy of doxycycline in treatment of early stages of mycosis fungoides (IA, IB and IIA) and to assess its apoptotic enhancing effect by studying the expression of BCL2 by the T lymphocytes.

Study Design

Randomized controlled trial

Population of study & disease condition

30 patients with early stage mycosis fungoides (Stage Ia,Ib and IIa)

Methodology in details

After signing an informed consent, each participant will be subjected to:

I. Baseline evaluation:

1. Baseline biopsy to document the current state of the disease and to assess immunohistochemically the expression of CD3 and Bcl2 by the lymphocytes.
2. Detailed history taking including onset, course, duration of the disease and history of any previous treatments used.
3. Detailed examination of skin lesions and scoring using:

   * Modified Severity of Index Weighted Assessment (mSWAT)
   * Composite Assessment of Index Lesion Severity (CAILS)
4. Pruritus scoring using a visual analog scale from 0-10, where 0=no pruritus and 10=worst imaginable pruritus
5. Photography

II. Treatment and dosing protocol:

Participants will be randomly allocated in either one of the treatment groups:

Group A: Will receive oral doxycycline in a dose of 200 mg daily for three months.

Group B: Will receive PUVA with dosing & increments according to the standard protocols of the Phototherapy Unit, Dermatology Department, Cairo University; 3 sessions per week for 3 months.

III. Timings of follow up visits and clinical assessments done:

Patients will be regularly assessed at weeks 4, 8, and 12. Patients continuing for another three months, as mentioned above, will be assessed at weeks 16, 20 and 24. The following will be done at these follow up visits: mSWAT, CAILS, pruritus scoring and photography. Side effects will be monitored and managed accordingly.

IV. Follow up biopsies:

A repeat biopsy will be taken at initial improvement in CAILS (or at week 12) for immunohistochemical re-assessment of the expression of CD3 and Bcl2 by the lymphocytes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (above 18) of either sex with established diagnosis of classic MF

Exclusion Criteria:

* Any variant of MF other than the classic variant.
* Advanced stages of classic MF: Stage IIb, III or IV.
* Pregnant and lactating females.
* Patients with autoimmune diseases e.g. SLE
* Patients with solid or hematological malignancies e.g. breast cancer, leukemia, etc.
* Patients with any contraindications for doxycycline (eg: liver disease, kidney disease, photosensitivity, peptic ulcer or patients receiving systemic retinoids).
* Patients with any contraindication to phototherapy (eg: any other skin cancers or photosensitivity); or to psoralen (eg: liver disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment | 3 months
  Clinical assessment of the extent of the lesions in body surface area

SECONDARY OUTCOMES:
Pathological assessment | 3months
  Pathological assessment using immunohistochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Mona AbdEl Halim, MD, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Dermatology departement, Cairo
  - Dermatology department, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valipour A, Jager M, Wu P, Schmitt J, Bunch C, Weberschock T. Interventions for mycosis fungoides. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD008946. doi: 10.1002/14651858.CD008946.pub3. PMID 32632956
- [Derived] El Sayed H, Shalaby S, Abdel-Halim MRE, Aboelfadl DM, Samir N. Efficacy of doxycycline in the treatment of early stages of mycosis fungoides: a randomized controlled trial. J Dermatolog Treat. 2021 Jun;32(4):424-431. doi: 10.1080/09546634.2019.1667474. Epub 2019 Sep 20. PMID 31526286